CLINICAL TRIAL: NCT02477085
Title: Methods of Labor Induction and Perinatal Outcomes : a Prospective National Study in France
Brief Title: Methods of Labor Induction and Perinatal Outcomes
Acronym: MEDIP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Nationale de sécurité du Médicament (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: AAP-2014-030
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Induction of Labor
Keywords: Labor; induction; delivery; prostaglandins; oxytocin; amniotomy; balloon catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all women with an induced labor: prospective population-based cohort of all women who have an induced labor during one month in seven perinatal networks
  Interventions: Other: all women with an induced labor

INTERVENTIONS:
Other: all women with an induced labor — all women who have an induced labor

SUMMARY:
Since it is a frequent intervention in Obstetrics, labor induction is rarely evaluated from national population-based cohorts. The study aims to assess the frequency of different induction methods used in France from a prospective population-based cohort of women with an induced labor. Maternal, fetal and neonatal outcomes will be compared between the different induction methods. Moreover the adhesion to national clinical guidelines concerning the induction of labor will be studied from this population-based cohort.

Finally the women satisfaction will be assessed according to the induction method used.

DETAILED DESCRIPTION:
Labor induction concerns about 22% of deliveries in France, according to the the 2010 French national perinatal survey. Labor induction could be associated with a higher risk of fetal and maternal complications, justifying its assessment from a population-based prospective cohort.

Several methods (dinoprostone, oxytocin, misoprostol, balloon catheter …) are used to induce labor in France. To decide and perform labor inductions, physicians can refer to published guidelines according to specific obstetrical situations. But many of these guidelines are based on a low level of evidence probably explaining observed differences in practices.

In some cases, labor induction is decided without indication, and women's involvement in this kind of decisions is not really evaluated.

The objectives are therefore :

* To evaluate the frequency of use of different methods for labor induction according to the cervix status, the indication of labor induction, and the place of the delivery.
* To analyse maternal, fetal and neonatal issues according to the different induction methods, taken into account the induction indications
* To compare current practices of labor induction to published national guidelines and to assess the impact of deviations from these guidelines on maternal and neonatal issues
* To assess women's satisfaction regarding the indication and the induction method used.

ELIGIBILITY:
Inclusion Criteria:

* patient who has a labor induction
* with a live fetus at the beginning of induction
* patient who did not have any opposition to use her medical and personal data or her child's medical data for research

Exclusion Criteria:

* in utero fetal death
* termination of pregnancy
* patient's refusal to participate to the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all women who have an induced labor
Sampling Method: Non-Probability Sample
Enrollment: 3049 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Composite measure of induction methods | Beginning of labor induction
  * Amniotomy
  * Amniotomy and oxytocin
  * Prostaglandins (PGE1, PGE2)
  * Balloon catheter
  For each of these methods, evaluation of these composite criteria
  * Frequency
  * Posology
  * Way of administration
  * Indication of labor induction

SECONDARY OUTCOMES:
Composite measure of maternal morbidity | Labor induction
  * Systemic infection
  * Uterine hyperkinesia
  * Uterine hypertonia
  * Instrumental delivery
  * Caesarean section
  * Degrees of perineal lacerations
  * Surgical complications
  * Uterine rupture
  * Manual removal of the placenta
  * Postpartum haemorrhage
  * Anaemia
  * Maternal transfer in ICU
Composite measure of fetal and neonatal mortality and morbidity | from induction up to average 7 days post delivery
  * Fetal heart rate anomalies during labor
  * Apgar score
  * Acidosis (pH < 7.10)
  * Intubation
  * Surfactant treatment administration
  * Non-invasive ventilation
  * Cardiopulmonary resuscitation
  * Adrenaline administration
  * Neonatal mortality
  * Neonatal trauma (fracture of long bones or skull, brachial plexus elongation, injury of the spinal cord, subdural hematoma)
  * Neonatal transfer in ICU
Women's satisfaction Questionnaire | 8 weeks after delivery
  18 questions about :
  * Woman's implication in the decision of labor induction
  * Woman's comprehension about the reason of labor induction
  * Woman's satisfaction about the decision/labor/delivery

CONTACTS AND LOCATIONS:
Overall Officials: Camille Le Ray, Principal Investigator — Assistance publique des Hôpitaux de Paris (APHP); François Goffinet, Study Director — Assistance publique des Hôpitaux de Paris (APHP)
Locations (1):
- Port-Royal maternity unit, Cochin Hospital, Assistance publique des Hôpitaux de Paris (APHP, Paris, France

REFERENCES:
- [Result] Jochum F, Le Ray C, Blanc-Petitjean P, Langer B, Meyer N, Severac F, Sananes N. Externally Validated Score to Predict Cesarean Delivery After Labor Induction With Cervi Ripening. Obstet Gynecol. 2019 Sep;134(3):502-510. doi: 10.1097/AOG.0000000000003405. PMID 31403585
- [Result] Blanc-Petitjean P, Schmitz T, Salome M, Goffinet F, Le Ray C; MEDIP Study Group. Target populations to reduce cesarean rates after induced labor: A national population-based cohort study. Acta Obstet Gynecol Scand. 2020 Mar;99(3):406-412. doi: 10.1111/aogs.13751. Epub 2019 Nov 19. PMID 31628852
- [Result] Blanc-Petitjean P, Salome M, Dupont C, Crenn-Hebert C, Gaudineau A, Perrotte F, Raynal P, Clouqueur E, Beucher G, Carbonne B, Goffinet F, Le Ray C. Labour induction practices in France: A population-based declarative survey in 94 maternity units. J Gynecol Obstet Hum Reprod. 2018 Feb;47(2):57-62. doi: 10.1016/j.jogoh.2017.11.006. Epub 2017 Nov 28. PMID 29196154